CLINICAL TRIAL: NCT03976544
Title: Natural Cycle Versus Hormone Replacement Therapy Cycle for a Frozen-thawed Embryo Transfer in PGT Patients: A Randomized Trial
Brief Title: Natural Cycle Versus Hormone Replacement Therapy Cycle for a Frozen-thawed Embryo Transfer in PGT Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: safety
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Caroline Roelens, Clinical fellow, CRG UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRT_NC-FET; 2018-003156-20 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Miscarriage; Frozen Embryo Transfer; Natural Cycle; Hormone Replacement Therapy Cycle; Preimplantation Genetic Screening; Euploid Embryos
Keywords: frozen-thawed embryo transfer; FET; natural cycle; hormone replacement therapy cycle; miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Estradiol; Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either natural cycle frozen-thawed embryo transfer (group A), or hormonal replacement therapy cycle frozen-thawed embryo transfer (group B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural cycle (No Intervention): Patients are asked to perform a blood sample, with evaluation of serum estradiol (E2), progesterone (P), luteinizing hormone (LH) and follicle stimulating hormone (FSH), on the first or second day of the menstrual cycle. If these serum hormonal values are considered basal for the beginning of the follicular phase, patients are asked to come back on day 10 to 12 of the cycle for blood sample and transvaginal ultrasound scan in order to assess follicular growth.
  The timing of ovulation is determined based on a combination of ultrasonography features (the presence of a dominant follicle and adequate endometrium) and endocrine hormonal values in serum blood samples. Ovulation is generally defined as an, at least, 180% increase of LH compared to the mean level in the previous 24h.
  Frozen-warmed blastocyst transfer will take place six days following the spontaneous LH surge.
- Hormone replacement therapy cycle (Experimental): Patients are asked to perform a blood sample, with evaluation of serum estradiol (E2), progesterone (P), luteinizing hormone (LH) and follicle stimulating hormone (FSH) on the first or second day of the menstrual cycle. If these values are considered basal for the beginning of the follicular phase, estrogen supplementation (Estradiol valerate, Progynova® 3x2mg/day) is started to induce proliferation of the endometrium. Blood sample and transvaginal ultrasound are thereafter performed ten to fourteen days later. If the endometrium is considered adequate (generally considered if triple line and above 6,5 mm thickness), embryo transfer is scheduled on the sixth day of progesterone (vaginal micronized progesterone, Utrogestan® 2x200mg twice a day) supplementation.
  In case of escape spontaneous ovulation embryo transfer will be performed considering the presumable time of ovulation.
  Interventions: Drug: Estradiol Valerate; Drug: Micronized progesterone

INTERVENTIONS:
Drug: Estradiol Valerate — Estradiol valerate will be started in the beginning of the menstrual cycle in order to induce proliferation of the endometrium.
  Other Names: Progynova
  Arms: Hormone replacement therapy cycle
Drug: Micronized progesterone — If the endometrium is considered adequately proliferated, micronized progesterone is administered and frozen-thawed blastocyst transfer will take place on the 6th day of supplementation.
  Other Names: Utrogestan
  Arms: Hormone replacement therapy cycle

SUMMARY:
The aim of the current study is to compare miscarriage rates (before 8 weeks) between a true natural cycle (awaiting spontaneous LH surge) and a hormone replacement therapy cycle prior to blastocyst transfer in preimplantation genetic testing (PGT) patients, with biopsy on day 5 of embryonic development. The advantage of performing the study in PGT patients is the exclusion of aneuploidy as a cause of miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* BMI under 35 kg/m2
* Regular menstrual cycle pattern (i.e. 24-35 days cycle)
* First, second and third ICSI-PGT cycle
* First frozen embryo transfer cycle following a fresh ICSI-PGT attempt
* PGT with trophectoderm biopsy on day 5 of embryonic development
* Signed informed consent

Exclusion Criteria:

* Oligo-amenorrhea
* BMI above 35
* Contraindications for the use of hormonal replacement therapy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 362 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Miscarriage rate before 8 weeks of gestation | 8 weeks
  a spontaneous loss of a clinical pregnancy before 8 weeks of gestational age, in which the embryo(s) is/are nonviable and is/are (not) spontaneously absorbed or expelled from the uterus per initiated embryo transfer cycle and per positive hCG

SECONDARY OUTCOMES:
Miscarriage rate after 8 weeks of gestation | 22 weeks
  a spontaneous loss of a clinical pregnancy after 8 weeks but before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus per initiated embryo transfer cycle and per positive hCG
Clinical pregnancy rate | 7 weeks
  a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy per initiated embryo transfer cycles
Ongoing pregnancy rate | 20 weeks
  the number of pregnancies after 20 weeks of gestation per initiated embryo transfer cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Reproductive Medicine UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03976544/Prot_000.pdf